CLINICAL TRIAL: NCT06343181
Title: A Qualitative Study on Treatment Adherence in Patients With Metastatic Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: IEO 1824
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Metastatic breast cancer (BC): Patients with diagnosis of BC

SUMMARY:
Qualitative observational study with the aim to explore medication adherence in a sample of patients with metastatic breast cancer.

Patients with metastatic breast cancer receiving or having received oral oncologic therapy, and attending the Division of Medical Senology at the European Institute of Oncology, will be included and enrolled in this research project."

DETAILED DESCRIPTION:
The aim of this research project is to assess the barriers and resources (both individual and environmental), as well as the psychological, clinical, and contextual factors that may influence adherence to pharmacological therapy in patients with actively treated metastatic breast cancer.

This will be achieved through a qualitative analysis focused on pharmacological therapy and its administration methods.

For this study, 4 focus groups will be conducted to identify the needs, barriers, and psychological, clinical, and contextual factors that may influence adherence to pharmacological treatment in patients with metastatic breast cancer, as well as their preferences regarding these treatments.

The number of focus groups was determined in accordance with recommendations from the literature for identifying relevant themes, which suggest that to achieve an adequate level of saturation, four or more focus groups are necessary.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old;
* Diagnosis of metastatic breast cancer;
* Availability of an internet connection and a PC or Tablet (for remote focus groups);
* Signing of the informed consent.

Exclusion Criteria:

* Presence of psychiatric or neurological conditions impairing the ability to comprehend the questions in Focus Groups or to express free consent to participate in the study;
* Presence of medical or oncological conditions other than metastatic breast cancer;
* Refusal to sign the informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of metastatic breast cancer treated at European Institute of Oncology
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of factors influencing patients' adherence to medical therapy | 1 month
  Collection of data in order to evaluation of factors influencing patient's adherence to medical treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella Pravettoni, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy